CLINICAL TRIAL: NCT04400409
Title: Implementation of Vascular Care Team to Improve Medical Management of Peripheral Arterial Disease (PAD) Patients
Brief Title: Implementation of Vascular Care Team to Improve Medical Management of PAD Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Colorado Prevention Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: OPTIMIZE PAD-1
Record Dates: First submitted 2020-05-19; First posted 2020-05-22 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Peripheral Artery Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Intervention A + site 6MWT administration (Active Comparator): Intervention A subjects will receive a vascular care team approach to care including pharmacy and healthcare provider assistance with medication adherence.
  6-Minute Walk Test (6MWT) will be administered by site staff.
  Interventions: Other: Intervention A - Vascular Care + site 6MWT administration
- Intervention B + site 6MWT administration (Active Comparator): Intervention B will receive standard care augmented with a single consultation with a Vascular Medicine physician who will provide the treating doctor with a personalized risk assessment for the patient and a summary of the 2018 American College of Cardiology (ACC)/American Heart Association (AHA) Guideline on Management of Blood.
  6-Minute Walk Test (6MWT) will be administered by site staff.
  Interventions: Other: Intervention B - Standard Care + site 6MWT administration
- Intervention A + CPC EQuIP 6MWT administration (Active Comparator): Intervention A subjects will receive a vascular care team approach to care including pharmacy and healthcare provider assistance with medication adherence.
  6-Minute Walk Test (6MWT) will be administered by CPC EQuIP staff.
  Interventions: Other: Intervention A - Vascular Care + CPC EQuIP 6MWT administration
- Intervention B + CPC EQuIP 6MWT administration (Active Comparator): Intervention B will receive standard care augmented with a single consultation with a Vascular Medicine physician who will provide the treating doctor with a personalized risk assessment for the patient and a summary of the 2018 American College of Cardiology (ACC)/American Heart Association (AHA) Guideline on Management of Blood.
  6-Minute Walk Test (6MWT) will be administered by CPC EQuIP staff.
  Interventions: Other: Intervention B - Standard Care + CPC EQuIP 6MWT administration

INTERVENTIONS:
Other: Intervention A - Vascular Care + site 6MWT administration — Implementation of multiple strategies related to improving lipid management, starting with a referral to the vascular care team. The subject will undergo a visit with a vascular care team, including a Vascular Medicine specialist who will obtain a patient history and prescribe a lipid lowering therapy regimen. The subject will also meet with a pharmacist to answer questions related to access to medications, drug side effects, and potential interactions with the subject's other medications. Additionally, the site staff will conduct and guide the subjects through 6MWTs at protocol-dictated time points.
  Arms: Intervention A + site 6MWT administration
Other: Intervention B - Standard Care + site 6MWT administration — Consists of provision of the treating provider with a copy of the 2018 ACC/AHA Guidelines on the Management of Blood Cholesterol. Subjects will return at 6 and 12 months for lab draws and endpoint event assessments but will not meet with vascular care team. Additionally, the site staff will conduct and guide the subjects through 6MWTs at protocol-dictated time points.
  Arms: Intervention B + site 6MWT administration
Other: Intervention A - Vascular Care + CPC EQuIP 6MWT administration — Implementation of multiple strategies related to improving lipid management, starting with a referral to the vascular care team. The subject will undergo a visit with a vascular care team, including a Vascular Medicine specialist who will obtain a patient history and prescribe a lipid lowering therapy regimen. The subject will also meet with a pharmacist to answer questions related to access to medications, drug side effects, and potential interactions with the subject's other medications. Additionally, the CPC EQuIP team will conduct and guide the subjects through 6MWTs at protocol-dictated time points.
  Arms: Intervention A + CPC EQuIP 6MWT administration
Other: Intervention B - Standard Care + CPC EQuIP 6MWT administration — Consists of provision of the treating provider with a copy of the 2018 ACC/AHA Guidelines on the Management of Blood Cholesterol. Subjects will return at 6 and 12 months for lab draws and endpoint event assessments but will not meet with vascular care team. Additionally, the CPC EQuIP team will conduct and guide the subjects through 6MWTs at protocol-dictated time points.
  Arms: Intervention B + CPC EQuIP 6MWT administration

SUMMARY:
This study intends to evaluate the efficacy of a multidisciplinary vascular care team utilizing an intensive guideline-based lipid reduction program in improving risk factor modification as measured by LDL-C reduction at 12 months in patients with peripheral artery disease (PAD). An additional objective is to understand the potential reach and impact if this program were extended across the University of Colorado Healthcare (UC Health) System.

DETAILED DESCRIPTION:
Patients with PAD and elevated LDL-C who are cared for at the University of Colorado (UC) and who provide consent will be randomized 1:1 to Intervention A, a vascular care team approach including pharmacy and healthcare provider assistance with medication adherence, versus Intervention B consisting of standard care augmented with a single consultation with a Vascular Medicine physician who will provide the treating doctor with a personalized risk assessment for the patient and a summary of the 2018 American College of Cardiology (ACC)/American Heart Association (AHA) Guideline on Management of Blood. In order to investigate the efficacy of the CPC Endpoint Quality Intervention Program (EQuIP), subjects will additionally be randomized 1:1 to an investigative site conducted Six-Minute Walk Test or an EQuIP team led Six-Minute Walk Test. Quality of Life data will be collected from all subjects. There will also be an observational cohort (registry) to understand current practice patterns and outcomes in a non-interventional PAD population within the UC Health system in order to assess the potential impact of Intervention A after conclusion of the randomized study.

ELIGIBILITY:
Inclusion Criteria:

1. Documented lower extremity atherosclerotic PAD with recommended goal LDL-C <70 mg/dL by the ACC/AHA Management of Blood Cholesterol Guidelines
2. Receiving care at CU Anschutz
3. Screening/baseline LDL-C ≥70 mg/dL without change in lipid lowering therapy within the last 30 days prior to LDL-C draw.
4. Able to provide informed consent and willing to participate

Exclusion Criteria:

1. Unwilling or unlikely to remain in the UC Health system through 1 year follow up (12 months after randomization)
2. Life expectancy < 12 months
3. Fasting triglycerides >400 mg/ml at screening
4. End-stage renal disease (eGRF<15 mL/min/1.73m2 and/or renal replacement therapy)
5. History of nephrotic syndrome
6. Clinical evidence of severe liver disease or another medical condition for which lipid lowering therapy may be contraindicated
7. Current enrollment in another investigational device or drug study with unapproved devices or therapies or with therapies that would impact lipid levels or lipid therapy
8. Any other condition that in the opinion of the investigator would make the subject unable to comply with the protocol

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2020-07-07 (Actual); Primary Completion 2023-05-11 (Actual); Study Completion 2023-05-11 (Actual)

PRIMARY OUTCOMES:
Month 12 LDL-C | 12 months
  Percent change from baseline to month 12 in LDL-C

SECONDARY OUTCOMES:
Month 6 LDL-C | 6 months
  Percent change from baseline at 6 months in LDL-C

OTHER OUTCOMES:
EQ-5D-5L Quality of Life questionnaire | 6 and 12 months
  Change from Baseline at months 6 and 12 in the EQ-5D-5L quality of life questionnaire.
Walking Impairment | 6 and 12 months
  Change from Baseline at months 6 and 12 in the Walking Impairment Questionnaire (WIQ)
Distance Walked | 6 and 12 months
  Change from Baseline at months 6 and 12 in the distance walked using the 6MWT.
Medication adherence | 6 and 12 months
  Proportions of subjects at months 6 and 12 adherent to lipid-lowering therapy, determined by self-reporting
Biomarker levels | 12 months
  Change from Baseline at 12 months in the levels of biomarkers (e.g. C-reactive protein [CRP], troponin, brain natriuretic peptide [BNP], lipoprotein(a) [Lp(a)])
Time to endpoint events | Time to event, up to 12 months
  Time from Baseline to:
  1. Major adverse cardiovascular events (MACE) (myocardial infarction [MI], ischemic stroke, or cardiovascular death) or major adverse limb event (MALE) (major amputation or acute limb ischemia);
  2. MACE
  3. MALE
  4. Lower extremity revascularization;
  5. Coronary artery revascularization;
  6. Death;
  7. Any hospitalization
Impact of CPC EQuIP process | 6 and 12 months
  Impact of CPC EQuIP process on variability in 6MWT at 6 and 12 months
Correlation between venipuncture and dried dried blood spots | 12 months
  Correlation between venipuncture and dried blood spot values of Baseline lipid and CRP levels

CONTACTS AND LOCATIONS:
Overall Officials: Connie Hess, MD, Principal Investigator — CPC Clinical Research
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Grundy SM, Stone NJ, Bailey AL, Beam C, Birtcher KK, Blumenthal RS, Braun LT, de Ferranti S, Faiella-Tommasino J, Forman DE, Goldberg R, Heidenreich PA, Hlatky MA, Jones DW, Lloyd-Jones D, Lopez-Pajares N, Ndumele CE, Orringer CE, Peralta CA, Saseen JJ, Smith SC Jr, Sperling L, Virani SS, Yeboah J. 2018 AHA/ACC/AACVPR/AAPA/ABC/ACPM/ADA/AGS/APhA/ASPC/NLA/PCNA Guideline on the Management of Blood Cholesterol: Executive Summary: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines. J Am Coll Cardiol. 2019 Jun 25;73(24):3168-3209. doi: 10.1016/j.jacc.2018.11.002. Epub 2018 Nov 10. No abstract available. PMID 30423391
- [Background] Bonaca MP, Nault P, Giugliano RP, Keech AC, Pineda AL, Kanevsky E, Kuder J, Murphy SA, Jukema JW, Lewis BS, Tokgozoglu L, Somaratne R, Sever PS, Pedersen TR, Sabatine MS. Low-Density Lipoprotein Cholesterol Lowering With Evolocumab and Outcomes in Patients With Peripheral Artery Disease: Insights From the FOURIER Trial (Further Cardiovascular Outcomes Research With PCSK9 Inhibition in Subjects With Elevated Risk). Circulation. 2018 Jan 23;137(4):338-350. doi: 10.1161/CIRCULATIONAHA.117.032235. Epub 2017 Nov 13. PMID 29133605
- [Background] Conte MS, Bandyk DF, Clowes AW, Moneta GL, Namini H, Seely L. Risk factors, medical therapies and perioperative events in limb salvage surgery: observations from the PREVENT III multicenter trial. J Vasc Surg. 2005 Sep;42(3):456-64; discussion 464-5. doi: 10.1016/j.jvs.2005.05.001. PMID 16171587
- [Background] Adam DJ, Beard JD, Cleveland T, Bell J, Bradbury AW, Forbes JF, Fowkes FG, Gillepsie I, Ruckley CV, Raab G, Storkey H; BASIL trial participants. Bypass versus angioplasty in severe ischaemia of the leg (BASIL): multicentre, randomised controlled trial. Lancet. 2005 Dec 3;366(9501):1925-34. doi: 10.1016/S0140-6736(05)67704-5. PMID 16325694
- [Background] Sabatine MS, Giugliano RP, Keech AC, Honarpour N, Wiviott SD, Murphy SA, Kuder JF, Wang H, Liu T, Wasserman SM, Sever PS, Pedersen TR; FOURIER Steering Committee and Investigators. Evolocumab and Clinical Outcomes in Patients with Cardiovascular Disease. N Engl J Med. 2017 May 4;376(18):1713-1722. doi: 10.1056/NEJMoa1615664. Epub 2017 Mar 17. PMID 28304224
- [Background] Bonaca MP, Braunwald E, Sabatine MS. Long-Term Use of Ticagrelor in Patients with Prior Myocardial Infarction. N Engl J Med. 2015 Sep 24;373(13):1274-5. doi: 10.1056/NEJMc1508692. No abstract available. PMID 26398078
- [Background] Arya S, Khakharia A, Binney ZO, DeMartino RR, Brewster LP, Goodney PP, Wilson PWF. Association of Statin Dose With Amputation and Survival in Patients With Peripheral Artery Disease. Circulation. 2018 Apr 3;137(14):1435-1446. doi: 10.1161/CIRCULATIONAHA.117.032361. Epub 2018 Jan 12. PMID 29330214
- [Background] Rehring TF, Stolcpart RS, Sandhoff BG, Merenich JA, Hollis HW Jr. Effect of a clinical pharmacy service on lipid control in patients with peripheral arterial disease. J Vasc Surg. 2006 Jun;43(6):1205-10. doi: 10.1016/j.jvs.2006.02.019. PMID 16765240